CLINICAL TRIAL: NCT01449864
Title: A Feasibility and Registration Study of Proton Radiotherapy for Upper Gastrointestinal Malignancies
Brief Title: Proton Radiotherapy for Upper Gastrointestinal Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 09211
Record Dates: First submitted 2011-10-07; First posted 2011-10-10 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Gastrointestinal Cancer
Keywords: upper GI malignancies; concurrent chemoradiation with continuous infusion 5-Fluorouracil chemotherapy
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton RT (Experimental): Subjects receive proton radiation
  Interventions: Radiation: Proton therapy

INTERVENTIONS:
Radiation: Proton therapy — The goal of radiation therapy is to deposit the majority of the radiation dose to the target while minimizing the dose to the surrounding normal tissues.

SUMMARY:
The primary objectives are to determine feasibility and the acute toxicity profile of proton therapy with concurrent continuous infusion 5-FU chemotherapy. Secondary objectives are to determine late toxicities and to generate preliminary data on clinical efficacy.

DETAILED DESCRIPTION:
This protocol invites patients with cancer of the upper digestive tract who will receive simultaneous proton radiation therapy and chemotherapy. The purpose of this study is to use a newer form of radiation therapy called proton radiation and to determine if its use is safe and effective in people with this type of cancer. Doctors will assess the safety of this method of treatment, record the side effects participants experience while receiving the standard dose of proton radiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic diagnosis of adenocarcinoma of the upper gastrointestinal tract, including patients with any of the following diagnoses and settings who are candidates to receive radiation which concurrent continuous infusion 5-FU chemotherapy: Pancreatic adenocarcinoma (unresected and adjuvant), Duodenal adenocarcinoma (unresected or adjuvant), Cholangiocarcinoma (unresected or adjuvant), Gastric adenocarcinoma (unresected or adjuvant), Gastroesophageal junction adeno carcinoma (adjuvant)
* Patient must be >18 years of age.
* Patient must have an ECOG Performance Status of 0-2, and a life expectancy of greater than or equal to 3 months.
* Patient must be able to provide informed consent.
* Women of child-bearing potential as long as she agrees to use a recognized method of birth control (e.g. oral contraceptive, IUD, condoms or other barrier methods etc.). Hysterectomy or menopause must be clinically documented.

Exclusion Criteria:

* Prior or simultaneous malignancies within the past two years (other than cutaneous squamous or basal cell carcinoma, melanoma in situ or thyroid carcinoma)
* Pregnant women, women planning to become pregnant and women that are nursing.
* Patients who experience surgical complications which prevent radiation from starting for 3 months or more.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Plastaras, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proton RT
Started | 22
Completed | 17
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Proton RT
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.79 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events
Description: Serious Adverse Events preventing more than 25% of planned treatments using proton radiotherapy.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Proton RT
Number analyzed (Participants) | 22
Participants | 0

2. Primary Outcome: Acute Toxicity
Description: Measured by experience of adverse events
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Proton RT
Number analyzed (Participants) | 22
Participants | 14

ADVERSE EVENTS:
Arm/Group | Proton RT
All-Cause Mortality (participants affected / at risk) | 5/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 15/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton RT (N=22)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (3)
Chills (General disorders) | 1 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Dermatitis radiation (Injury, poisoning and procedural complications) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dizziness (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 6 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Floaters (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 3 (5)
Pain (General disorders) | 1 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes